CLINICAL TRIAL: NCT04659655
Title: VIenna Pilot Study for Automated Annular Suturing Technology to Assist in Aortic & Mitral Valve Replacement - A Single-center Clinical Safety & Feasibility Pilot Trial
Brief Title: VIenna Pilot Study for Automated Annular Suturing Technology
Acronym: VIP-RAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: LSI SOLUTIONS, Inc. (Unknown)
Responsible Party: Principal Investigator, Martin Andreas, M.D., Assoc. Prof. PD MD MBA, PhD, MEBCTS, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC 1660/2019
Record Dates: First submitted 2020-11-16; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Aortic Valve Disease; Mitral Valve Disease
Keywords: surgical aortic valve replacement; surgical mitral valve replacement
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- surgical aortic valve replacement (Other): n=20 patients with aortic valve pathology and indication for surgical aortic valve replacement
  Interventions: Procedure: automated annular suturing
- surgical mitral valve replacement (Other): n=10 patients with mitral valve pathology and indication for surgical mitral valve replacement
  Interventions: Procedure: automated annular suturing

INTERVENTIONS:
Procedure: automated annular suturing — RAM® Automated Suturing Technology. The RAM® DEVICE and SEW-EASY® DEVICE are automated suturing devices indicated for use in the approximation of soft tissue and prosthetic materials when used in conjunction with RAM® COR-SUTURE® QUICK LOAD® surgical suture. Devices will be used for the approximation of respective replacement valves during surgical aortic or mitral valve replacement as described in the study protocol. Cases may include use of the RAM® RING/RAM® RACK devices for suture management and the Aortic Root Retractor (ARR) with delivery device.

SUMMARY:
The objective of this study is to compare surgical outcomes between patients who underwent valve replacement with and without the help of the automated annular suturing technology. In addition, data of the early and intermediate postoperative period will be collected within routine clinical follow-up in order to assess morbidity and mortality as well as echocardiographic parameters.

DETAILED DESCRIPTION:
This study is a clinical, single-center pilot-study to evaluate safety and performance. 30 Patients (n=20 aortic valve replacement/ n=10 mitral valve replacement) with aortic and mitral valve pathology, highly likely for prosthetic valve replacement, who are planned for surgery at the Vienna General Hospital (AKH) will be included in this study with respect to the inclusion and exclusion criteria. The patients will undergo aortic or prosthetic mitral valve replacement using a specified automated annular suturing system for placement of the annular pledgeted sutures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low to moderate operative risk (Defined by STS mortality risk below 8%)
* Patients above the age of 18 years
* Patients willing and able to sign the informed consent

Exclusion Criteria:

* Patients with active endocarditis
* Patients with previous cardiac surgery other than pacemaker implantation
* Emergency procedures
* Patient who did not sign the informed consent form and/ or refuse to participate
* Patients unable to read or understand the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from mortality at 30 days post-OP assessed by clinical follow-up reports. | 30 days post surgical valve replacement
  Follow-ups 30 days post-OP are performed and freedom from mortality evaluated.
Implantation time assessed by surgical report. | procedural
  Implantation time, the duration defined from start of the valve assessment until the completion of the prosthesis implantation (defined as fixation of the last suture) assessed by surgical report.

SECONDARY OUTCOMES:
Freedom from severe adverse events at 30 days post-OP assessed by clinical follow-up reports | 30 days post surgical valve replacement
  Follow-ups 30 days post-OP are performed to and freedom from severe adverse events evaluated.
Surgical times assessed by surgical report. | procedural
  Surgical times, aortic cross-clamp time and cardiopulmonary-bypass time, assessed by surgical report.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Andreas, Assoc. Prof. PD MD MBA, PhD,, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong JK, Melvin AL, Siordia JA, Joshi DJ, Sauer JS, Knight PA. Novel Automated Suturing Technology for Minimally Invasive Aortic Valve Replacements. Ann Thorac Surg. 2018 Feb;105(2):645-649. doi: 10.1016/j.athoracsur.2017.07.054. Epub 2017 Nov 27. PMID 29174775
- [Background] Johnson CA Jr, Melvin AL, Lebow BF, Yap A, Knight PA. Video assisted right mini-thoracotomy for aortic valve replacement. J Vis Surg. 2018 Feb 27;4:39. doi: 10.21037/jovs.2018.01.16. eCollection 2018. PMID 29552521
- [Background] Robinson DA, Sagebin F, Yap AJ, Johnson CA Jr, Knight PA. Aortic valve replacement with annular enlargement via a right anterior minithoracotomy. Multimed Man Cardiothorac Surg. 2018 Jul 26;2018. doi: 10.1510/mmcts.2018.044. PMID 30070778
- [Background] Nellis JR, Fitch ZW, Choi AY, Meza JM, Spector ZZ, Von Bergen NH, Torres JE, Klapper JA, Sauer JS, Turek JW. A Minimally Invasive Approach for Placing Sew-On Epicardial Leads in the Child. Innovations (Phila). 2018 Nov/Dec;13(6):455-457. doi: 10.1097/IMI.0000000000000568. PMID 30540590
- See also: LSI SOLUTIONS, Inc. — https://www.lsisolutions.com/